CLINICAL TRIAL: NCT02618811
Title: Enhanced Recovery After Surgery Protocol (ERAS) in Colorectal Surgery Diminishes the Negative Impact of Sarcopenia on Short Term Outcomes
Brief Title: ERAS in Colorectal Surgery Diminishes the Negative Impact of Sarcopenia on Short Term Outcomes
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Michał Pędziwiatr, MD PhD, Jagiellonian University
Other Study IDs: JagiellonianU-03
Record Dates: First submitted 2015-11-22; First posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Sarcopenia; Colonic Neoplasms
Keywords: sarcopenia; myosteatosis; enhanced recovery after surgery; colorectal cancer; minimally invasive surgery; complications
MeSH Terms: conditions — Sarcopenia; Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: not sarcopenic
- Group 2: sarcopenic
- Group 3: not myosteatotic
- Group 4: myosteatotic

SUMMARY:
So far, the impact of sarcopenia has been analysed only in patients undergoing traditional surgical procedures (laparotomy) or those with metastatic spread. As the ERAS protocol combined with minimally invasive access decreases postoperative metabolic disorders, it seems possible that it can limit the deleterious impact of sarcopenia as well. The aim of this study was to investigate whether the use of ERAS protocol in colorectal cancer patients influences the postoperative risk due to sarcopenia.

DETAILED DESCRIPTION:
The prospective observation with post-hoc analysis of 171 consecutive colorectal cancer patients was performed. In all patients 16-item ERAS protocol was applied.

Contrast-enhanced CT scan was performed preoperatively. From each scan one CT image at the level of L3 vertebra was transferred in Digital Imaging and Communications in Medicine format (DICOM) and anonymised. Firstly, the threshold range between -29 and +150 Hounsfield units was set to semi-automatically outline muscle areas, - 150 to - 50 was used for visceral adipose tissue areas, and -190 to -30 was used for subcutaneous and intermuscular adipose tissue areas. Secondly, the software calculated the surface area (cm2) of each tissue. The L3 skeletal muscle area (rectus abdominis, external and internal obliques, transversus abdominis, quadratus lumborum, psoas, erector spinae) normalized for patient height was used to calculate skeletal muscle index (SMI) (cm2/m2).

According to Martin et al. sarcopenia was defined as a SMI <41 cm2/m2 in women, <43 cm2/m2 in men with a BMI <25 kg/m2, and <53 cm2/m2 in men with a BMI >25 kg/m2 (10). To assess for myosteatosis the mean radiodensity of a L3 psoas muscle was measured. The cut-off for patients with BMI <25 kg/m2 was <41 Hounsfield units and <33 Hounsfield units for patients with BMI ≥25 kg/m2.

For the purposes of further analysis the entire group of patients was divided into subgroups depending on the presence of sarcopenia or myosteatosis.

ELIGIBILITY:
Inclusion Criteria:

* confirmed adenocarcinoma of colon or rectum
* complete preoperative radiology assessment with abdominal CT scan
* laparoscopic resection
* perioperative care according to ERAS principles

Exclusion Criteria:

* unavailability of a preoperative abdominal CT scan (within 30 days prior surgery)
* emergency or initially open surgery
* patients treated with endoscopic techniques: transanal endoscopic microsurgery (TEM), transanal total mesorectal excision (TaTME)
* concomitant inflammatory bowel diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analysis included prospectively collected data from consecutive patients electively operated for colorectal cancer in the years 2014-2015. All patients were operated using laparoscopic surgery, and the perioperative care was based on pre-established ERAS protocol consisting of 13 items
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Complications | up to 30 days post surgery

SECONDARY OUTCOMES:
Hospital length of stay (days) | up to discharge from hospital, an average 6 days
Compliance with ERAS protocol (%) | up to discharge from hospital, an average 6 days
Tolerance of oral diet on the 1st postoperative day | up to discharge from hospital, an average 6 days
  tolerating at least 800 ml of clear water/fluids and 1 oral nutritional supplement within the first 24h postoperative hours
Time to first flatus | up to discharge from hospital, an average 6 days
Readmission rate | up to 30 days post surgery
Mobilization on the 1st postoperative day | up to discharge from hospital, an average 6 days
  walking at least 100 m without assistance, at least 6h out of bed (sitting, walking)
Need for opioid analgesia postoperatively | up to discharge from hospital, an average 6 days
  no need for opioid drug administration (any kind, dosage or administration route)

CONTACTS AND LOCATIONS:
Overall Officials: Michał Pędziwiatr, MD, PhD, Principal Investigator — 2nd Department of Surgery, Jagiellonian University, Krakow, Poland
Locations (1):
- 2nd Department of General Surgery, Jagiellonian University, Krakow, Poland

REFERENCES:
- [Background] Greco M, Capretti G, Beretta L, Gemma M, Pecorelli N, Braga M. Enhanced recovery program in colorectal surgery: a meta-analysis of randomized controlled trials. World J Surg. 2014 Jun;38(6):1531-41. doi: 10.1007/s00268-013-2416-8. PMID 24368573
- [Background] Vlug MS, Wind J, Hollmann MW, Ubbink DT, Cense HA, Engel AF, Gerhards MF, van Wagensveld BA, van der Zaag ES, van Geloven AA, Sprangers MA, Cuesta MA, Bemelman WA; LAFA study group. Laparoscopy in combination with fast track multimodal management is the best perioperative strategy in patients undergoing colonic surgery: a randomized clinical trial (LAFA-study). Ann Surg. 2011 Dec;254(6):868-75. doi: 10.1097/SLA.0b013e31821fd1ce. PMID 21597360
- [Background] Huang DD, Wang SL, Zhuang CL, Zheng BS, Lu JX, Chen FF, Zhou CJ, Shen X, Yu Z. Sarcopenia, as defined by low muscle mass, strength and physical performance, predicts complications after surgery for colorectal cancer. Colorectal Dis. 2015 Nov;17(11):O256-64. doi: 10.1111/codi.13067. PMID 26194849
- [Background] Jones KI, Doleman B, Scott S, Lund JN, Williams JP. Simple psoas cross-sectional area measurement is a quick and easy method to assess sarcopenia and predicts major surgical complications. Colorectal Dis. 2015 Jan;17(1):O20-6. doi: 10.1111/codi.12805. PMID 25328119
- [Background] Thoresen L, Frykholm G, Lydersen S, Ulveland H, Baracos V, Prado CM, Birdsell L, Falkmer U. Nutritional status, cachexia and survival in patients with advanced colorectal carcinoma. Different assessment criteria for nutritional status provide unequal results. Clin Nutr. 2013 Feb;32(1):65-72. doi: 10.1016/j.clnu.2012.05.009. Epub 2012 Jun 12. PMID 22695408
- [Background] Martin L, Birdsell L, Macdonald N, Reiman T, Clandinin MT, McCargar LJ, Murphy R, Ghosh S, Sawyer MB, Baracos VE. Cancer cachexia in the age of obesity: skeletal muscle depletion is a powerful prognostic factor, independent of body mass index. J Clin Oncol. 2013 Apr 20;31(12):1539-47. doi: 10.1200/JCO.2012.45.2722. Epub 2013 Mar 25. PMID 23530101
- [Background] Malietzis G, Aziz O, Bagnall NM, Johns N, Fearon KC, Jenkins JT. The role of body composition evaluation by computerized tomography in determining colorectal cancer treatment outcomes: a systematic review. Eur J Surg Oncol. 2015 Feb;41(2):186-96. doi: 10.1016/j.ejso.2014.10.056. Epub 2014 Nov 3. PMID 25468746